CLINICAL TRIAL: NCT07046117
Title: Effect of Tezepelumab on Barrier Function in Severe Asthmatic Patients With and Without Comorbid Chronic Rhinosinusitis With Nasal Polyps - an Exploratory Study
Brief Title: Effect of Tezepelumab on Barrier Function in Severe Asthmatic Patients With and Without Comorbid Chronic Rhinosinusitis With Nasal Polyps
Acronym: Tezebarrier
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marco Idzko, Univ.Prof.Dr.med., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Tezebarrier2025
Record Dates: First submitted 2025-06-05; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Asthma Bronchiale; Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Keywords: asthma; chronic rhinosinusitis with nasal polyps; tezepelumab; epithelial barrier; airways
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma only (Active Comparator): Patients suffering from asthma in absence of CRSwNP will be administerd tezepelumab every 4 weeks
  Interventions: Drug: Tezepelumab
- Asthma with CRSwNP (Active Comparator): Patients suffering from Asthma with CRSwNP will be administered Tezepelumab every 4 weeks
  Interventions: Drug: Tezepelumab

INTERVENTIONS:
Drug: Tezepelumab — injection with Tezepelumab every 4 weeks

SUMMARY:
In this study, we will investigate the effect of tezepelumab on the epithelial barrier function of the upper and lower airways in patients suffering from severe asthma with and without chronic rhinosinusitis with nasal polyps. This will be achieved by analysis of epithelial barrier function upon challenge with various harmful substances (e.g. cigarette smoke extract, allergens) in cultured primary respiratory tract epithelial cells. Furthermore we will assess changes in clinical parameters, cellular composition and inflammatory mediators.

DETAILED DESCRIPTION:
The primary objective of the proposal is to investigate the effect of Tezepelumab on the epithelial barrier function of upper and lower airways. To that aim, epithelial cells from the upper and lower airways will be cultured to investigate the change in barrier function during Tezepelumab treatment in patients suffering from severe asthma in presence or absence of chronic rhinosinusitis with nasal polyps. In addition, mucus plugging will be quantified by computer tomography before and after Tezepelumab therapy. These data will be supplemented by cellular and mediator analyses as well as microbiome analyses. Thus, our study will unravel the molecular mechanisms and benefits underlying therapy with Tezepelumab in patients suffering from severe asthma with or without nasal polyps.

Objectives Primary objective: Effect of Tezepelumab treatment on the barrier function of upper and lower airways in patients suffering from severe asthma with and without CRSwNP. This will be achieved by analysis of epithelial barrier function upon challenge with various harmful substances (e.g. cigarette smoke extract, allergens, and rhinovirus) in cultured primary respiratory tract epithelial cells using the xCELLigence system for continuous monitoring of barrier function.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Age 18-99 years and willing to participate in the study
3. Have a recorded clinical diagnosis of asthma (ICD-10 Code: J45)
4. Undergo severe asthma treatment according to GINA/DAL treatment step 4 or 5
5. Meet the requirements for treatment of severe asthma with Tezepelumab defined as:

   * severe asthma that remains uncontrolled despite a high dosage of ICS/LABA, or that requires a high dose to prevent it from becoming uncontrolled. One of the following criteria needs to be fulfilled:

     * ACT <20, ACQ>0.75
     * During the last 12 months 2 courses of OCS for at least 3 days due to severe asthma symptoms
     * During last 12 months one exacerbation requiring hospitalization
     * Lung function: FEV1 <80% predicted
   * FeNO ≥ 20 ppB
   * had either ≥250 eosinophils /µl measured in the blood OR measurement of blood eosinophils ≥150 cells during reduction of OCS dosing or high dose ICS and/or one measurement of sputum eosinophils > 2% or BAL eosinophils > 2%
   * Group with polyps: Presence of nasal polyps as confirmed by endoscopy or CT according to the European Position Paper on Rhinosinusitis and Nasal Polyps Guidelines
6. mucus score of ≥ 1
7. Patients with a history of treatment with monoclonal antibodies for asthma or polyps will only be included if at least a washout period of 3 half-lives or 3 months have passed (whichever is longer)

Exclusion Criteria:

* 1. Patients with current therapy with biologics as well as therapy with biologics 12 weeks (3 half-lives) before the start of the study or history of therapy with tezepelumab 2. Pregnancy (as determined by urine pregnancy test) 3. Patients with severe anatomic variations or deviations that do not allow access to all areas in the nasal cavity or to perform bronchoscopy 4. Patients with any other confounding underlying lung disorder including but not limited to:

  * Bronchiectasis, pulmonary fibrosis, emphysema, primary ciliary dyskinesia
  * Cystic fibrosis, any known parasitic infections and lung cancer

    5. Patients with other causes of nasal polyps than Type 2 CRS inflammation 6. Patients with pulmonary conditions with symptoms of asthma and blood eosinophilia including but not limited to: Eosinophilic granulomatosis with polyangiitis (EGPA) allergic bronchopulmonary aspergillus and hypereosinophilic syndrome 7. Contraindications for endobronchial and/or transbronchial biopsy. 8. A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study 9. Patients with clinically meaningful comorbidity as determined by the evaluating committee 10. Immunosuppressive treatment (e.g. cyclosporine) 11. Drug and alcohol abuse 12. Current smoker and former smokers if stopped smoking <6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in cell index | 6 months
  Changes in normalized cell index in response to barrier-damaging substances in cultured primary epithelial cells of the different disease entities using the xCELLigence system for continuous monitoring of barrier function.

SECONDARY OUTCOMES:
Change in mucus plugging | 6 months
  The extent of air-trapping, bronchial wall thickening and mucus plugging per pulmonary segment will be scored independently by two thoracic radiologists.
Change in marker expression immune cell subsets | 6 months
  Cellular composition and marker expression on cells derived from Bronchoalveolar lavage (BAL), nasal polyps and blood as assessed by a multi-colour mass cytometry panel
Change in inflammatory mediators | 6 months
  (Inflammatory) mediator expression in BAL, lung tissue, nasal mucosa, polyp tissue (e.g. OLINK explorer)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Idzko, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes
Scientific Data will be shared in public available databases
Supporting Information: Analytic Code
Time Frame: from Dec 2025 with open end
Access Criteria: those who are registerd with public databases or who contact the investigators via email